CLINICAL TRIAL: NCT04381767
Title: EYE-SYNC Concussion Classification Study
Status: Completed | Type: Observational
Sponsor: Sync-Think, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EYESYNCCCV2020
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Concussion, Mild; Concussion; Eye; Concussion, Brain; Concussion, Severe; Brain Injuries; Concussion, Cerebral
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Concussion Evaluation: Adult athletes receiving a clinical evaluation for a suspected concussion after head injury
  Interventions: Device: EYE-SYNC

INTERVENTIONS:
Device: EYE-SYNC — Evaluation of oculomotor performance using visual presentation and eye tracking analysis
  Other Names: SCAT-5

SUMMARY:
The purpose of this study is to determine the sensitivity and specificity of an aid in assessment of concussion based on eye-tracking, in comparison to a clinical reference standard appropriate for sport-related concussion evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women actively engaged in competitive athletics
* Eye tracking measurements and SCAT5 evaluations are collected within 3-day window
* Eye tracking measurements and SCAT5 evaluations are collected within 3 days of injury

Exclusion Criteria:

* Prior enrollment (subjects may only enroll once)
* POOR eye tracking data quality
* Subjects without reported injury detailing alteration of consciousness (AOC) or altered mental status (AMS) defined as self-report, witness report or the following responses to the SCAT5 SSS: "Difficulty Remembering" ≥ 4 or "Confusion" ≥ 4, or scored less than 23 on the SCAT5 Standardized Assessment of Concussion (SAC) or greater than 25 on the SCAT5 Symptom Severity Score (SSS)
* EYE-SYNC smooth pursuit standard deviation of tangential error (SDTE) variance scores < 2.0

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include all patients evaluated for potential traumatic brain injury presenting to the sports medicine clinicians in an athletic environment.
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
A change in metrics of eye movement that enable positive concussion detection using EYE-SYNC metrics | 3 days
  A True Positive and True Negative rate for identifying Concussion as compared to a Clinical Reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Sync-Think, Inc., Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No